CLINICAL TRIAL: NCT02868125
Title: Radiography Protocol in the Acute Phase After Proximal Femur Internal Fixation- Self Assessment and Recommendations
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, David segal, MD, Dr. David Segal, Meir Medical Center
Other Study IDs: 0172
Record Dates: First submitted 2016-08-10; First posted 2016-08-16 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-08

CONDITIONS: Pertrochanteric Fracture
Keywords: pertrochanteric; radiography
MeSH Terms: interventions — Portable X-Ray

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Radiation: X ray radiography — All studied patients will undergo an x-ray radiography of the operated hip. This protocol is a part of the investigators' common practice policy regardless of the study.

SUMMARY:
There is no standardized protocol regarding the post-operative radiographic follow up of patients that sustain pertrochanteric hip fractures and are treated with closed reduction and internal fixation. The policy in the investigator's institution as in other hospitals is to conduct a radiogram of the operated hip during the first days following operation after the patient bore weight on the fixated femur. The investigator's goal is to asses the added value of this policy and to offer recommendations regarding this specific followup component.

DETAILED DESCRIPTION:
There is no consensus regarding the proper radiographic protocol following closed reduction and internal fixation of pertrochanteric femoral fractures. Despite its' questionable necessity and significant economic burden, many medical centers practice a policy of imaging internally fixated proximal femurs after the patients bore weight on them. The investigator's goal is to assess the added value of the postoperative imaging study described.

Materials and methods: We will conduct a prospective study. All patients who will be treated with closed reduction and internal fixation of AO31A fractures will be enrolled. Two sets of imaging studies will be assessed- the intra-operative AP and axial fluoroscopy studies and the radiograms that are taken following bearing weight on the operated hip. Three decision steps will take place regarding weight bearing limitations and a necessity for re-operation- (1) Immediately after the operation; (2) A day after the operation; (3) Following weight bearing according to a new radiogram. Objective measurements will be taken for each hip on both imaging modalities- neck-shaft angle, neck length and tip-apex distance.

ELIGIBILITY:
Inclusion Criteria:

* Pertrochanteric femur fracture, classified as AO-31-A
* Go through a closed reduction and internal fixation operation at the investigator's institution

Exclusion Criteria:

* patients that due to clinical findings or other necessities go through specific followup radiography imaging protocols
* Fluoroscopy imaging studies were not saved

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients of all ages who sustain a pertrochanteric femur fracture, classified as AO-31-A, and go through a closed reduction and internal fixation operation at the investigator's institution.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2016-05; Primary Completion 2017-05 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Changes in weight bearing instructions on follow up x ray imaging | OIne week
  During the few day following surgery a decision has to be made regarding weight bearing limitations on the operated hip. patients can be instructed to: (1) Full weight bearing, (2) Partial weight bearing, (3) Touch-down weight bearing, (4) Non weight bearing. This decision is primary taken according to the intra-operative fluoroscopy images, and revised a few days later after examining the first follow up x-ray imaging of the operated hip. The investigators wish to learn whether a new data from the first follow up imaging study leads to changes in weight bearing instructions. If a change was made due to new findings on follow up x-ray, then the case would be regarded as "change", while if no changes were made they would be regarded as "no change". Finally the investigators will calculate the number of patients that need to go through follow up x-ray imaging studies in order for one patient to have their weight bearing instructions changed.

SECONDARY OUTCOMES:
Changes in neck shaft angle between intra-operative fluoroscopy and follow-up x ray imaging studies | one week
  Neck-shaft angle is the angle between the femoral neck and femoral shaft, measured in degrees. The investigators wish to find whether there is a difference in the measurements' outcome for the same patients on intra-operative fluoroscopy and on the first post-operative followup x-ray imaging studies. The angle described will be calculated on both modalities and compared, with the outcome being the difference in degrees.
The need for reoperation | One week
  During the few day following surgery a decision has to be made regarding need for re-operation. This decision is primary taken according to the intra-operative fluoroscopy images, and revised a few days later after examining the first follow up x-ray imaging of the operated hip. The decision is based on both objective features such as nec-shaft angle, tip-apex index and neck length, and on subjective features such as the patients' basic medical functional status. The investigators wish to learn whether a new data from the first follow up imaging study leads to changes in the decision for re-operation. If a change was made due to new findings on follow up x-ray, then the case would be regarded as "change", while if no changes were made they would be regarded as "no change". Finally the investigators will calculate the number of patients that need to go through follow up x-ray imaging studies in order for one patient to be advised differently for re-operation.
Changes in neck length between intra-operative fluoroscopy and follow-up x ray imaging studies | One week
  Neck length is the distance between the femoral neck base and the femoral head, and is measured in millimeters. The investigators wish to find whether there is a difference in the measurement outcome for the same patients on intra-operative fluoroscopy and on the first post-operative followup x-ray imaging studies. The length described will be calculated on both modalities and compared, with the outcome being the difference in millimeters.
Changes in tip-apex distance between intra-operative fluoroscopy and follow-up x ray imaging studies | One week
  Tip apex distance is the sum of the distances measured on both AP and axial studies between the proximal lag screw tip and the proximal femoral head border . It is measured by millimeters. The investigators wish to find whether there is a difference in the measurement outcome for the same patients on intra-operative fluoroscopy and on the first post-operative followup x-ray imaging studies. The length described will be calculated on both modalities and compared, with the outcome being the difference in millimeters.

CONTACTS AND LOCATIONS:
Overall Officials: David Segal, MD, Principal Investigator — Meir Medical Center
Locations (1):
- Meir Medical Center, Kfar Saba, Israel

IPD SHARING:
Plan to Share IPD: No
no data will be shared

REFERENCES:
- [Background] Tufescu T. Working toward reducing postoperative fracture radiographs: a survey of Canadian surgeons. Can J Surg. 2016 Feb;59(1):26-8. doi: 10.1503/cjs.005715. PMID 26812405
- [Background] van Embden D, Stollenwerck GA, Koster LA, Kaptein BL, Nelissen RG, Schipper IB. The stability of fixation of proximal femoral fractures: a radiostereometric analysis. Bone Joint J. 2015 Mar;97-B(3):391-7. doi: 10.1302/0301-620X.97B3.35077. PMID 25737524
- [Derived] Segal D, Palmanovich E, Faour A, Marom E, Feldman V, Yaacobi E, Slevin O, Kish B, Brin YS. Routine early post-operative X-ray following internal fixation of intertrochanteric femoral fractures is unjustified: a quality improvement study. J Orthop Surg Res. 2018 Jul 31;13(1):189. doi: 10.1186/s13018-018-0896-9. PMID 30064462